CLINICAL TRIAL: NCT05062031
Title: Comparison of Defocus Incorporated Multiple Segments® (DIMS®) Lenses Alone Versus Monofocal Lenses + Atropine 0.05% Eyedrops on the Evolution of Ocular Axial Length at 2 Years in Myopia Control in Children: Single-centre Prospective Randomised Controlled 1:1 Open-label Non-inferiority Study
Brief Title: Myopia Control in Children: Comparison of Defocus Incorporated Multiple Segments® Lenses Versus Atropine 0.05% Eyedrops
Acronym: ATROSMART
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: Ecouter Voir (Unknown); Hoya Lens France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMN_2021_11
Record Dates: First submitted 2021-09-09; First posted 2021-09-30 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Myopia
Keywords: Myopia; Pediatric ophthalmology; Myopia control; Defocus Incorporated Multiple Segments (DIMS) lenses; Low concentration atropine
MeSH Terms: conditions — Myopia | interventions — Lenses; Atropine; Ophthalmic Solutions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DIMS® (Experimental): Defocus Incorporated Multiple Segments® lenses
  Interventions: Device: Defocus Incorporated Multiple Segments® (DIMS®) lenses
- Low-concentration atropine + monofocal lenses (Active Comparator)
  Interventions: Drug: Atropine 0.05% eyedrops; Device: Monofocal lenses

INTERVENTIONS:
Device: Defocus Incorporated Multiple Segments® (DIMS®) lenses — Daily wear for 24 months. Lenses have a central monofocal optical zone correcting spherical or spherocylindrical ametropia, surrounded by a ring made up of 300 defocusing pellets. This lens geometry reduces the phenomenon of blurred image projected in the retinal periphery, encountered when myopic eyes are corrected with monofocal lenses.
  Other Names: Miyosmart®
  Arms: DIMS®
Drug: Atropine 0.05% eyedrops — One drop each evening in both eyes for 24 months.
  Other Names: Low-concentration atropine
  Arms: Low-concentration atropine + monofocal lenses
Device: Monofocal lenses — Daily wear for 24 months
  Arms: Low-concentration atropine + monofocal lenses

SUMMARY:
Myopia is the most common refractive disorder in the world. Many strategies have been developed to control myopia in children. Among them, the instillation of low-concentration atropine eyedrops has been proven to be effective in numerous publications. Nevertheless, the spreading of atropine use is limited by: (1) its uneven availability, (2) a proportion of children with no or poor response, (3) some issues of long-term compliance (4) the possibility of a rebound effect after treatment cessation.

Among the non-drug myopia control strategies, corrective lenses including the Defocus Incorporated Multiple Segments® (DIMS®) technology have demonstrated their effectiveness in a previous study (Hong Kong) when compared to monofocal lenses.

The aim of this study is to compare the efficacy of DIMS lenses alone versus atropine 0.05% eyedrops + monofocal lenses, on the evolution of ocular axial length at 2 years in myopic children.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of myopia - measured under cycloplegia - defined by:

  1. A sphere power between -1 and -6 Diopters, on at least one of the two eyes
  2. AND a cylindrical power strictly inferior to 2 Diopters
  3. AND a maximum refractive error strictly inferior to 8 Diopters in the flattest axis
* Not benefiting and never having benefited from a myopia control strategy (orthokeratology, soft defocusing lenses, low concentration atropine eye drops, peripheral defocusing corrective lenses)
* Written consent of both parents

Exclusion Criteria:

* History of genetic disease, or general condition suggesting a syndromic myopia (including an axial length greater than 27 mm)
* Strabismus
* Amblyopia defined by a best corrected visual acuity strictly inferior to 10/10 on one of the two eyes
* Anisometropia defined by a difference of 2 Diopters or more between the two eyes (in spherical equivalent)
* History of allergy to atropine
* History of severe anaphylaxis
* Optical correction with contact lenses
* Previous ophthalmologic surgery of the cornea, lens, retina
* History of glaucoma or any other chronic ophthalmological disease in the course of treatment (including vernal keratoconjunctivitis)

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 242 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Axial length measurements | Inclusion, 24 months
  Difference between the mean of 6 axial length measurements (in mm) acquired with the IOLMaster 500® at 24 months and the mean of 6 axial length measurements at inclusion
Spherical equivalent | Pre inclusion (screening consultation in the 15 days preceding inclusion), 24 months
  Difference in spherical equivalent (in diopters) under cycloplegia on autorefractometer at 24 months and at preinclusion

CONTACTS AND LOCATIONS:
Overall Officials: Gilles MARTIN, MD, Principal Investigator — Hôpital Fondation Adolphe de Rothschild
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, France